CLINICAL TRIAL: NCT02375334
Title: Comparative Development of Data Driven Systems for Insuring Timely Monitoring for Brain Tumor Patients for Management of Myelosuppression
Brief Title: Adherence Monitoring System in Managing Myelosuppression in Patients With Newly Diagnosed Malignant Gliomas Receiving Temozolomide and Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Support Staff Left Institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00013273; NCI-2015-00113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99115; CCCWFU # 99115 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-02-11; First posted 2015-03-02 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Malignant Glioma; Myelosuppression
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical chart review): Patient lab and visit dates are monitored by the Cancer Center ORIS and EPIC based systems during the 42 days of the concurrent temozolomide and radiation therapy.
  Interventions: Other: Medical Chart Review

INTERVENTIONS:
Other: Medical Chart Review — Medical chart review by the Cancer Center ORIS and EPIC based systems
  Other Names: Chart Review

SUMMARY:
This research trial studies an adherence monitoring system in managing myelosuppression in patients with newly diagnosed malignant gliomas who are receiving temozolomide and radiation therapy. The development of an adherence monitoring system may help doctors more effectively utilize electronic medical records to manage myelosuppression during standard treatment with temozolomide and radiation therapy in patients with malignant gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop an adherence monitoring system within Epic that is functionally equivalent to the previously designed and validated system in the Cancer Center Oncology Research Information System (ORIS) for patients with newly diagnosed malignant gliomas receiving concurrent temozolomide and radiation therapy.

II. To test the newly designed Epic system by comparing the frequency and timing of flags (laboratory date flags, visit date flags and in-patient status flags) and non-adherent days generated with the frequency and timing of those generated by ORIS for patients with newly diagnosed malignant gliomas receiving concurrent temozolomide and radiation therapy.

SECONDARY OBJECTIVES:

I. To develop both systems so that they may be easily adapted in the future to other therapies that require compliance monitoring.

OUTLINE:

Patient lab and visit dates are monitored by the Cancer Center ORIS and EPIC based systems during the 42 days of the concurrent temozolomide and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive concurrent temozolomide and radiation therapy for newly diagnosed malignant gliomas during and after the construction of the system until the end of the study

Exclusion Criteria:

* Patients participating in clinical trials or other deviations from standard therapies that engender similar monitoring risk will be evaluated for this study on a case by case basis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive concurrent temozolomide and radiation therapy for newly diagnosed malignant gliomas
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Development of a new adherence monitoring system within Epic that is functionally equivalent to the previously designed and validated system in the Cancer Center ORIS | 42 days
  To compare the two systems, the McNemar's tests of paired proportions will be used to compare the output of the established software system to the new system built into the EMR reporting structure.
Frequency and timing of flags (laboratory date flags, visit date flags and in-patient status flags) generated with the new system | 42 days
  To compare the two systems, the McNemar's tests of paired proportions will be used. For each day, whether or not any flag (laboratory date flags, visit date flags and in-patient status flags) was generated or whether a gap occurred will be characterized. By day, the two systems will be compared to determine if they agree for flags and gap days (separately). Alternative methods will be used (such as conditional logistic regression with a random subject effect) if correlation between days is observed.
Non-adherent days generated with the new system | 42 Days
  To compare the two systems, the McNemar's tests of paired proportions will be used. For each day, whether or not any flag (laboratory date flags, visit date flags and in-patient status flags) was generated or whether a gap occurred will be characterized. By day, the two systems will be compared to determine if they agree for flags and gap days (separately). Alternative methods will be used (such as conditional logistic regression with a random subject effect) if correlation between days is observed.

SECONDARY OUTCOMES:
Expansion of both systems to other therapies that require compliance monitoring | 42 days
  The feasibility of expanding the systems scope to other disease/treatment scenarios that require compliance monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States